CLINICAL TRIAL: NCT05615181
Title: Evaluation of the French Translation of Gothenburg Trismus Questionnaire (GTQ)
Acronym: TRISMUS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-06
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Trismus
Keywords: trismus; Patient reported outcomes; u Gothenburg Trismus Questionnaire
MeSH Terms: conditions — Trismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A monocentric Study to evaluate the french translation of Gothenburg Trismus Questionnaire (GTQ).

DETAILED DESCRIPTION:
Trismus is defined as a limitation in the mouth/jaw-opening ability due to a reduced mandible mobility. Trismus can occur from benign jaw related conditions, often referred to as temporomandibular disorders (TMD). It can also result from local or metastatic tumor growth of head and neck (H&N) tumors, and more importantly, as a debilitating side-effect to H&N oncology treatment, especially radiotherapy

The Gothenburg Trismus Questionnaire (GTQ) is a Patient Reported Outcome, validated in English, portuguese and sweden language.

The aim of this study is to develop a new tool in french language and to evaluate the specific impact of trismus on quality of life .

ELIGIBILITY:
* Inclusion Criteria:

  * Patient treated for trismus
  * Age ≥ 18 years old
  * Read, write and understand the French language
* Exclusion Criteria:

  * Patient under guardianship, deprived of liberty, safeguard of justice
  * Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated for trismus
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Gothenburg Trismus Questionnaire (GTQ) | once at inclusion
  patient Reported Outcome measure: score 0-4 (0 means a better outcome, 4 means a worse outcome.)

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Valence, Valence, Drome, France

IPD SHARING:
Plan to Share IPD: Undecided